CLINICAL TRIAL: NCT05852951
Title: Cycle and Ovulation Study Expansion
Status: Completed | Type: Observational
Sponsor: Apple Inc. (Industry)
Collaborators: Exponent (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00054031
Record Dates: First submitted 2023-03-07; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Menstruation
Keywords: menstruation; ovulation; menstrual cycle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Menstrual patterns: Regular menstrual cycles and irregular menstrual cycles; irregular menstrual cycles are defined as having variation in menstrual cycles of greater than 2 days and less than 2 months

SUMMARY:
The objective of this study was to collect menstrual cycle, health sensor data and general health information to understand correlations between menstrual cycle and health sensor data, and how those correlations may be affected by general health. Participants entered menstrual cycle information (such as start dates, end dates, symptoms, flow), basal body temperature as measured by a thermometer, and ovulation and progesterone test results via apps installed on their iPhone. Additionally, participants were provided with an Apple Watch and a wrist-worn hardware prototype wrist-worn sleep band to collect physiological sensor data. Both menstrual cycle information and physiological sensor data stored on the participants' iPhone prior to enrolling in the study (up to 18 months) was also collected. This study aimed to collect data from females aged 14 and older who are currently menstruating with irregular and regular menstrual cycles.

ELIGIBILITY:
* At least 14 years of age (19 for residents of Alabama and Nebraska and 21 for residents of Mississippi)
* Can communicate in written and spoken English
* Own functioning iPhone iOS 14 or later, with access to reliable data plan and Wifi
* Access to reliable Wifi in the bedroom
* Willingness to participate in remote visits and follow study procedures for the duration of the study, including use of Apple Watch and a wrist-work hardware prototype
* Able to read and understand the written consent form
* Reside in the US for the duration of the study

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Contract research organization
Sampling Method: Non-Probability Sample
Enrollment: 698 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Retrospective ovulation day estimate | 12 months
  Retrospective ovulation day estimation (algorithm uses multiple measurements including menstrual flow, urine ovulation prediction testing, basal body temperature, overnight aggregated wrist temperature)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Qing, PhD, Principal Investigator — Exponent
Locations (1):
- Exponent, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Park J, Zhang CY, Jukic AMZ, Baird DD, Coull BA, Hauser R, Mahalingaiah S, Zhang S, Curry CL. Performance of algorithms using wrist temperature for retrospective ovulation day estimate and next menses start day prediction: a prospective cohort study. Hum Reprod. 2025 Mar 1;40(3):469-478. doi: 10.1093/humrep/deaf005. PMID 39881571